CLINICAL TRIAL: NCT05975294
Title: Prospective Comparative Study Between Ultrasound-guided Continuous Erector Spinae Plane Block and the Use of Intravenous Patient Controlled Analgesia for Management of Pain in Patients With Multiple Fracture Ribs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Azmy, assistant lecteurer anaethesia and ICU department sohag univerisity hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-07-01MD
Record Dates: First submitted 2023-07-27; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Multiple Fracture Ribs
MeSH Terms: interventions — Fentanyl; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group(E): (Active Comparator): including 30 patients with multiple fracture ribs will undergo ultrasound guided continuous erector spinae plane block with abolus 0.3ml /kg of amixture 0.125% bupivicaine with fentanyl of 2 mic per ml then Infusion of 0.1 ml /kg/hr of the same mixture.
  Interventions: Drug: amixture 0.125% bupivicaine with fentanyl
- Group (C) (Active Comparator): including 30 patients with multiple fracture ribs will be given intravenous PCA device of 100 ml volume containing 80 mg of nalbuphine ,180 mg ketorolac, 24mg dexamethasone, 16 mg danset and normal saline at a rate of 2 ml/h.
  Interventions: Drug: 100 ml volume containing 80 mg of nalbuphine ,180 mg ketorolac, 24mg dexamethasone, 16 mg danset

INTERVENTIONS:
Drug: amixture 0.125% bupivicaine with fentanyl — ultrasound guided continuous erector spinae plane block with abolus 0.3ml /kg of amixture 0.125% bupivicaine with fentanyl of 2 mic per ml then Infusion of 0.1 ml /kg/hr of the same mixture.
  Arms: Group(E):
Drug: 100 ml volume containing 80 mg of nalbuphine ,180 mg ketorolac, 24mg dexamethasone, 16 mg danset — PCA device of 100 ml volume containing 80 mg of nalbuphine ,180 mg ketorolac, 24mg dexamethasone, 16 mg danset and normal saline at a rate of 2 ml/h.
  Arms: Group (C)

SUMMARY:
Rib fractures are common after blunt injury to the chest. Present in 10% of blunt trauma admissions. Pain associated with rib fractures can result in compromise of pulmonary function causing hypoxaemia or pneumonia, which may require mechanical ventilation. Adequate relief of rib fracture pain allows the patient to breathe deeply, avoid intubation and clear secretions effectively, which will minimise the pulmonary complications .

Pain control is essential for not only primary pain relief but also preventing secondary complications such as atelectasis or pneumonia as well as the transition to chronic pain. Accordingly, further steps are now being taken from the conventional pain control medication and techniques by the introduction of more aggressive pain control measures .Traditional regional anaesthesia (RA) techniques such as paravertebral, intercostal and epidurals injections are resource-intensive and time-consuming, limited to single dermatomes; provide incomplete analgesia of the hemithorax; and are associated with significant potential complications such as local anaesthetic intoxication, vasovagal syncope, hemi diaphragmatic paresis and pneumothorax .

The erector spinae plane block (ESPB) is a novel fascial plane block. Its use has been documented in numerous instances with positive outcomes in controlling acute as well as chronic pain. The most popular technique was the continuous infusion through a catheter . Fascial plane blocks that can be used for rib fracture pain management are serratus anterior plane block, erector spinae plane block and the rhomboid intercostal and subserratus (RISS) block. The procedure is more simple to use with a lower incidence of complications ,less time consuming , more superficial than others so it can be used in patients on anticoagulant therapy .

Providing analgesia for patients with rib fractures continues to be a management challenge. Therefore, further studies are needed comparing between different techniques to prove their efficacy in pain management

ELIGIBILITY:
Inclusion Criteria:

* • Age 18:60 years

  * Patient with 2 or more unilateral rib fractures.
  * ASA 1 , ASA 2

Exclusion Criteria:

* • patient refusal

  * History of chronic pain or daily use of analgesics
  * History of psychiatric disorder or inability to understand the consent form or how to use a visual analog scale (VAS) for pain measurement
  * Severe renal or hepatic dysfunction
  * Allergy to any required drug
  * Second thoracic surgery
  * Local infection at the injection site
  * Spinal deformity
  * head injury
  * lung complications related to trauma ( pneumothorax , haemothorax , lung collapse).
  * need of mechanical ventilation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
• Pulmonary function to evaluate mean change in incentive spirometry volume | 1 year
  from pretreatment then 1 h after procedure then daily for 5days including: Forced expiratory volume in one second (FEV1) ,Forced vial capaciy (FVC) and The ratio of the two volumes(FEV1/FVC) and inspiratory capacity (IC).
• VAS pain score | 1 year
  will be calculated pretreatment then at 0, 0.5h, 1h, 2h , 3h ,6h, 12h and 24h thn daily for 5 days at rest and at movement.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Truitt MS, Murry J, Amos J, Lorenzo M, Mangram A, Dunn E, Moore EE. Continuous intercostal nerve blockade for rib fractures: ready for primetime? J Trauma. 2011 Dec;71(6):1548-52; discussion 1552. doi: 10.1097/TA.0b013e31823c96e0. PMID 22182865
- [Background] Kumar G, Kumar Bhoi S, Sinha TP, Paul S. Erector spinae plane block for multiple rib fracture done by an Emergency Physician: A case series. Australas J Ultrasound Med. 2020 Aug 30;24(1):58-62. doi: 10.1002/ajum.12225. eCollection 2021 Feb. PMID 34760612
- [Background] Hwang EG, Lee Y. Effectiveness of intercostal nerve block for management of pain in rib fracture patients. J Exerc Rehabil. 2014 Aug 31;10(4):241-4. doi: 10.12965/jer.140137. eCollection 2014 Aug. PMID 25210700
- [Background] Picard J, Meek T. Complications of regional anaesthesia. Anaesthesia. 2010 Apr;65 Suppl 1:105-15. doi: 10.1111/j.1365-2044.2009.06205.x. PMID 20377552